CLINICAL TRIAL: NCT03856411
Title: A Phase III, Randomized, Double-blind, Placebo-controlled, Multi-center Clinical Study to Evaluate the Efficacy and Safety of Toripalimab Injection (JS001) or Placebo Combined With First-line Standard Chemotherapy in Treatment-naive Advanced Non-small Cell Lung Cancer (NSCLC)
Brief Title: A Study to Evaluate the Efficacy and Safety of Toripalimab or Placebo Combined With Chemotherapy in Treatment-naive Advanced NSCLC
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Shanghai Junshi Bioscience Co., Ltd. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: JS001-019-III-NSCLC
Record Dates: First submitted 2019-01-24; First posted 2019-02-27 (Actual); Last update posted 2023-02-01 (Actual); Status verified 2023-01

CONDITIONS: Treatment-naive Advanced Non-small Cell Lung Cancer
MeSH Terms: interventions — toripalimab; Drug Therapy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group TORIPALIMAB combined with standard chemotherapy (Experimental)
  Interventions: Drug: TORIPALIMAB INJECTION (JS001 ) combine with chemotherapy
- Group Placebo combined with standard chemotherapy (Placebo Comparator)
  Interventions: Drug: TORIPALIMAB INJECTION (JS001 ) combine with chemotherapy

INTERVENTIONS:
Drug: TORIPALIMAB INJECTION (JS001 ) combine with chemotherapy — TORIPALIMAB INJECTION(JS001 ) or Placebo ,240mg/6ml/vial, Q3W,up to 2 years of treatment.
  Other Names: JS001, TAB001

SUMMARY:
This is one randomized, double-blind, placebo-controlled, multi-center, phase III clinical study to evaluate the efficacy and safety of Toripalimab injection (JS001) or placebo combined with standard 1st-line chemotherapy in treatment-naïve advanced non-small cell lung cancer (NSCLC); and evaluate the population with the best predictive biomarkers, i.e., positive diagnosis population.

About 450 subjects with advanced non-small cell lung cancer without activated EGFR mutation (exon 19 deletion, or exon 21 L858R, exon 21 L861Q, exon 18 G719X or exon 20 S768I mutations) and ALK fusion will be 2:1 randomized into two groups, JS001 combined with the standard 1st-line chemotherapy will be given in the study group whereas placebo combined with standard 1st-line chemotherapy will be given in the control group. The stratification will be based on the following factors:

PD-L1 expression (TC≥1% vs TC<1%); Smoking state (often smoking vs no smoking or infrequent smoking); Pathological type (squamous cell carcinoma vs non-squamous cell carcinoma).

ELIGIBILITY:
Inclusion Criteria:

Only the patients meeting all the following criteria can be eligible to participate in the trial:

1. Histologically and/or cytologically confirmed stage IV non-small cell lung cancer and ALK fusion
2. At least one measurable lesion 3 No history of any systemic anti-tumor therapy.

4. Agreement on providing formalin fixed tumor tissue specimen or fresh biopsy tissue from tumor lesions after diagnosis of metastasis 6. Age of 18-75 years 7. ECOG Scores 0-1; 8. Expected survival ≥ 3 months;

Exclusion Criteria:

1. Known allergy to recombinant humanized anti-PD-1 monoclonal antibody drug and its components;
2. Histologically or cytopathologically confirmed combination with small cell lung cancer component or sarcomatoid lesion;
3. Current participation in and receiving other study treatment, or participation in treatment of one study drug within 4 weeks prior to administration of JS001;
4. Previous use of systematic chemotherapy for advanced NSCLC; targeted therapy for advanced NSCLC
5. Previous use of anti-PD-1 antibody, anti-PD-L1 antibody, anti-PD-L2 antibody or anti-CTLA-4 antibody (or any other antibody acting on T cells synergetic stimulation or checkpoint pathway, such as IDO, IL-2R, GITR);
6. Chest (lung) radiotherapy > 30 Gy within 6 months prior to the start of study treatment.
7. Active tuberculosis (TB), receiving anti-tuberculosis therapy currently or within one year prior to screening;
8. Known active central nervous system (CNS) metastasis and/or cancerous meningitis;
9. Spinal cord compression for which operation and/or radical radiotherapy has not been given, or no clinical evidence of stable disease for ≥4 weeks prior to enrollment after treatment for previously diagnosed spinal cord compression
10. Uncontrolled pleural effusion, pericardial effusion, or ascites requiring repeated drainage
11. Uncontrollable or symptomatic hypercalcemia
12. Clinically uncontrolled active infection, including but not limited to acute pneumonia;
13. Uncontrollable major epileptic seizure or superior vena cava syndrome
14. Previous or current combination with other malignancies ;
15. History of idiopathic pulmonary fibrosis, organized pneumonia (e.g., obliterating bronchiolitis), drug induced pneumonia, idiopathic pneumonia or evidence of active pneumonia during chest CT scanning for screening;
16. Known hepatic diseases of clinical significance, including active viral hepatitis, alcoholic hepatitis or other hepatitis, liver cirrhosis, fatty liver, hereditary liver disease;
17. Use of systemic immunosuppressive therapy for any active autoimmune disease within two years prior to Day 1 of the 1st cycle;
18. Vaccination of live-virus vaccine within 30 days after the start of planned treatment

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 465 (Actual)
Dates: Start 2019-03-18 (Actual); Primary Completion 2022-08-31 (Actual); Study Completion 2023-01-09 (Actual)

PRIMARY OUTCOMES:
PFS | Up to 2 approximately years
  Progression free survival (PFS) evaluated by investigators according to the response evaluation criteria in solid tumors (RECIST 1.1)

SECONDARY OUTCOMES:
OS | Up to 2 approximately years
  Overall survival (OS)
PFS | Up to 2 approximately years
  PFS evaluated by the Blinded Individual Review Committee (BIRC) based on RECIST1.1 criteria
ORR | Up to 2 approximately years
  Objective response rate (ORR) evaluated by investigators and BIRC based on RECIST1.1
DOR | Up to 2 approximately years
  Duration of response (DOR) evaluated by investigators and BIRC based on RECIST1.1
DCR | Up to 2 approximately years
  Disease control rate (DCR) evaluated by investigators and BIRC based on RECIST1.1
TTR | Up to 2 approximately years
  Time to response (TTR) evaluated by investigators and BIRC based on RECIST1.1
Incidence of AEs/SAEs | From date of consent informed until 60 days after the last investigational product administration. Up to 2 approximately years
  Overall incidence of adverse events (AEs); incidence of grade 3 and above AEs; incidence of serious adverse events (SAEs); incidence of AEs leading to termination of the investigational drug; incidence of AEs interruption of the investigational drug

CONTACTS AND LOCATIONS:
Locations (1):
- Cancer Hospital Chinese Academy of Medical Sciences, Beijing, Beijing Municipality, China

REFERENCES:
- [Derived] Zhong J, Fei K, Wu L, Li B, Wang Z, Cheng Y, Li X, Wang X, Han L, Wu X, Fan Y, Yu Y, Lv D, Shi J, Huang J, Zhou S, Han B, Sun G, Guo Q, Ji Y, Zhu X, Hu S, Zhang W, Wang Q, Jia Y, Wang Z, Song Y, Wu J, Shi M, Li X, Han Z, Liu Y, Yu Z, Liu AW, Wang X, Zhou C, Zhong D, Miao L, Zhang Z, Zhao H, Yang J, Wang D, Wang Y, Li Q, Zhang X, Ji M, Yang Z, Cui J, Gao B, Wang B, Liu H, Nie L, He M, Jin S, Gu W, Shu Y, Zhou T, Feng J, Yang X, Huang C, Zhu B, Yao Y, Yao S, Yu J, Cai SL, Cai Y, Xu J, Zhuang W, Luo X, Duan J, Wang J. Toripalimab plus chemotherapy for first line treatment of advanced non-small cell lung cancer (CHOICE-01): final OS and biomarker exploration of a randomized, double-blind, phase 3 trial. Signal Transduct Target Ther. 2024 Dec 24;9(1):369. doi: 10.1038/s41392-024-02087-6. PMID 39715755
- [Derived] Zhao J, Wang L, Zhou A, Wen S, Fang W, Zhang L, Duan J, Bai H, Zhong J, Wan R, Sun B, Zhuang W, Lin Y, He D, Cui L, Wang Z, Wang J. Decision model for durable clinical benefit from front- or late-line immunotherapy alone or with chemotherapy in non-small cell lung cancer. Med. 2024 Aug 9;5(8):981-997.e4. doi: 10.1016/j.medj.2024.04.011. Epub 2024 May 22. PMID 38781965
- [Derived] Zhang M, Xu K, Lin Y, Zhou C, Bao Y, Zhang L, Li X. Cost-effectiveness analysis of toripalimab plus chemotherapy versus chemotherapy alone for advanced non-small cell lung cancer in China. Front Immunol. 2023 May 29;14:1169752. doi: 10.3389/fimmu.2023.1169752. eCollection 2023. PMID 37313403
- [Derived] Wang Z, Wu L, Li B, Cheng Y, Li X, Wang X, Han L, Wu X, Fan Y, Yu Y, Lv D, Shi J, Huang J, Zhou S, Han B, Sun G, Guo Q, Ji Y, Zhu X, Hu S, Zhang W, Wang Q, Jia Y, Wang Z, Song Y, Wu J, Shi M, Li X, Han Z, Liu Y, Yu Z, Liu AW, Wang X, Zhou C, Zhong D, Miao L, Zhang Z, Zhao H, Yang J, Wang D, Wang Y, Li Q, Zhang X, Ji M, Yang Z, Cui J, Gao B, Wang B, Liu H, Nie L, He M, Jin S, Gu W, Shu Y, Zhou T, Feng J, Yang X, Huang C, Zhu B, Yao Y, Tang X, Yu J, Maher E, Feng H, Yao S, Keegan P, Wang J. Toripalimab Plus Chemotherapy for Patients With Treatment-Naive Advanced Non-Small-Cell Lung Cancer: A Multicenter Randomized Phase III Trial (CHOICE-01). J Clin Oncol. 2023 Jan 20;41(3):651-663. doi: 10.1200/JCO.22.00727. Epub 2022 Oct 7. PMID 36206498